CLINICAL TRIAL: NCT01479920
Title: The Identification of Central Neural Network for Antidepressant Effects of Dense Cranial Electroacupuncture Stimulation - a Positron Emission Topographic (PET) Study
Brief Title: A Positron Emission Topographic (PET) Study on Depression Patient With Electroacupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Kowloon Hospital, Hong Kong (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 09-091
Record Dates: First submitted 2011-11-16; First posted 2011-11-28 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Depressive Disorder; Depressive Symptoms; Depressive Syndrome; Emotional Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCEAS (Active Comparator): Dense cranial electroacupuncture stimulation (DCEAS)
  For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Interventions: Drug: Fluoxetine; Procedure: DCEAS (Hwato®/ Dongbang®)
- n-CEA (Sham Comparator): Non-invasive cranial electroacupuncture (n-CEA)
  For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Interventions: Drug: Fluoxetine; Procedure: n-CEA (Strietberger®)

INTERVENTIONS:
Drug: Fluoxetine — Subjects of both study arms received orally administered SSRIs for 4 weeks in an open manner. For those who were currently under antidepressant treatment, they would continue the existing treatment regimens. For those who were not medicated at the time of trial, fluoxetine (FLX) was given at an initiate dose of 10 mg/day and escalated to an optimal dose within one week, based on individual response, but the maximum dose was set at 40 mg/day.
  Other Names: Prozac; Sarafem; Fontex; Zactin; Lovan; Fluohexal; Auscap; Depreks; Floxet; Flunil; Fluox; Fluzac; Fluxen
Procedure: DCEAS (Hwato®/ Dongbang®) — Six pairs of cranial acupoints are used: Baihui (Du-20) and Yintang (EX-HN3), left Sishencong (EX-HN1) and Toulinqi (GB15), right Sishencong (EX-HN1) and Toulinqi (GB15), bilateral Shuaigu (GB8), bilateral Taiyang (EX-HN5), and bilateral Touwei (ST8). All these acupoints are located on the forehead.
  Disposable acupuncture needles (Hwato®/ Dongbang®, 0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm obliquely into acupoints, on which low- and high-frequency alternating electrical stimulation with continuous waves is conducted for 30 min. The intensity is adjusted to a level at which patients feel comfortable.
  Other Names: Hwato®; Dongbang®
  Arms: DCEAS
Procedure: n-CEA (Strietberger®) — Streitberger's acupuncture needles will be applied on the same acupoints, with the same electrical stimulation parameters, except that the needles only adhere to the skin instead of insertion.
  Other Names: Strietberger®
  Arms: n-CEA

SUMMARY:
This is a randomized, assessor-blind, placebo controlled study in major depressive disorder (MDD) patients. Subjects receiving antidepressant drug (FLX) would be assigned to receive either 18 sham / active DCEAS for in 6 weeks. Changes in the severity of depressive symptoms over time are measured using depression rating scales. Brain glucose metabolic levels are measured using PET at baseline and endpoint. The most intriguing and expected result might be that acupuncture treated-patients may display comparable or even better outcomes and the clinical improvements by acupuncture are correlated with the restoration of the activities in the related brain regions.

DETAILED DESCRIPTION:
Although the development of various classes of antidepressant drugs, represented by selective serotonin reuptake inhibitors (SSRI), has considerably improved the prognosis and the tolerability in the treatment of depressive disorders, the currently available antidepressant therapy is still incomplete, because there are about 40% of depressed individuals who cannot obtain full response and a large proportion of the patients experience recurrent episodes.

Recently the principal investigator has completed a clinical trial to test whether dense cranial electroacupuncture stimulation (DCEAS) could enhance the antidepressant efficacy in the early phase of SSRI treatment (fluoxetine, FLX) of major depressive disorder (MDD). It was found that DCEAS is clinically safe and effective in augmenting the antidepressant efficacy in early SSRI treatment. As we hypothesize that this normalizing effect is associated with the modulation of various nervous functions associated with the pathophysiology of MDD, we design this neuroimaging (PET) DCEAS study to delineate the related mechanisms.

The objective of this study are:

1) To compare clinical improvements on depressive symptoms between DCEAS and FLX monotherapy in MDD subjects; (2) To determine the effects of DCEAS treatment on glucose metabolic levels in related brain regions in comparison with healthy controls and FLX-treated patients, using PET scanning; and (3) To correlate between clinical improvements and changes in PET-measured activities of related brain regions in a pool of the subjects treated with DCEAS and FLX.

In this 6-week, assessor-blind, randomized, controlled study of DCEAS as additional treatment with the antidepressant drug FLX, a total of 82 patients with major depressive disorder (MDD) will be recruited. The patients will be randomly assigned to FLX (10-30 mg/day) combined with sham (n =41) or FLX with active DCEAS (n =41) (18 sessions, 3 sessions a week). Changes in the severity of depressive symptoms over time are measured using depressive instruments. Clinical response and remission rates are also calculated. Two sessions of PET scan will be conducted at baseline and endpoint. The study will be conducted at HKU School of Chinese Medicine, Queen Mary Hospital, and Kowloon Hospital, Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. with righthandedness;
2. have first-episode MDD diagnosed as the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV); and
3. HAMD-17 score is ≥ 20; and
4. never had any psychoactive medications.

Exclusion Criteria:

1. unstable medical conditions;
2. have suicidal ideas or attempts or aggressive behavior;
3. previously experienced manic, hypomanic, or mixed episode;
4. immediate family members have bipolar or psychotic disorders;
5. treatment with investigational drugs in past 6 months;
6. alcoholism or drug abuse in past 1 year; or
7. have needle phobia.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
HAMD-17 | 42-day (course of treatment)
  Depression symptoms is measured using the 17-item Hamilton Depression Scale. Assessments will be conducted at baseline and once weekly thereafter.
SDS | 42-day (course of treatment)
  Depression symptoms is measured using the Self-Rating Depression Scale (SDS). Assessments will be conducted at baseline and once weekly thereafter.

SECONDARY OUTCOMES:
PET scanning | 42-day (course of treatment)
  The secondary outcome measure of high interest is the results of PET scanning. Two sessions of PET scan will be conducted at baseline and endpoint for enrolled subjects. An additional group of age- and gender-matched healthy subjects will be invited for one-session PET scan.
Clinical response | 42-day (course of treatment)
  Clinical response, defined as greater than or equal to 50% reduction at endpoint from baseline on HAMD-17, is measured at the baseline and once weekly thereafter.
Remission | 42-day (course of treatment)
  Remission, defined as 7 points or less on HAMD-17 score, is measured at the baseline and once weekly thereafter.
Latency | 42-day (course of treatment)
  The latency of the clinical response.
Adverse events | 42-day (course of treatment)
  Adverse events are assessed using the Treatment Emergent Symptom Scale (TESS) when applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (4):
- China (3):
  - School of Traditional Chinese Medicine, Southern Medical University, Guangzhou
  - Department of Psychiatry, Queen Mary Hospital, Hong Kong
  - Department of Psychiatry, Kowloon Hospital, Kowloon
- Department of Diagnostic Radiology, The University of Hong Kong, Hong Kong, Hong Kong